CLINICAL TRIAL: NCT01231607
Title: A Study of the Efficacy and Safety of Multiple Doses of Dutasteride Versus Placebo and Finasteride in the Treatment of Male Subjects With Androgenetic Alopecia
Brief Title: Dutasteride Versus Placebo and Finasteride in Men With Androgenetic Alopecia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 114263
Record Dates: First submitted 2010-10-28; First posted 2010-11-01 (Estimated); Results first posted 2012-10-04 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-06

CONDITIONS: Androgenetic Alopecia
MeSH Terms: conditions — Alopecia | interventions — Dutasteride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1mg Finasteride (Active Comparator): 1mg finasteride active plus dutasteride placebo, by mouth once daily
  Interventions: Drug: 1mg Finasteride active; Drug: Dutasteride placebo
- 0.02mg Dutasteride (Active Comparator): 0.02mg dutasteride active plus finasteride placebo, by mouth once daily
  Interventions: Drug: 0.02mg dutasteride; Drug: Finasteride placebo
- 0.1mg Dutasteride (Active Comparator): 0.1mg dutasteride active plus finasteride placebo, by mouth once daily
  Interventions: Drug: 0.1mg dutasteride; Drug: Finasteride placebo
- 0.5mg Dutasteride (Active Comparator): 0.5mg dutasteride active plus finasteride placebo, by mouth once daily
  Interventions: Drug: 0.5mg dutasteride; Drug: Finasteride placebo
- Placebo (Placebo Comparator): 1mg finasteride placebo plus dutasteride placebo, by mouth once daily
  Interventions: Drug: Finasteride placebo; Drug: Dutasteride placebo

INTERVENTIONS:
Drug: 1mg Finasteride active — 1mg finasteride active, by mouth once daily
  Arms: 1mg Finasteride
Drug: 0.02mg dutasteride — 0.02mg dutasteride active, by mouth once daily
  Arms: 0.02mg Dutasteride
Drug: 0.1mg dutasteride — 0.1mg dutasteride active, by mouth once daily
  Arms: 0.1mg Dutasteride
Drug: 0.5mg dutasteride — 0.5mg dutasteride active, by mouth once daily
  Arms: 0.5mg Dutasteride
Drug: Finasteride placebo — finasteride placebo, by mouth once daily
  Arms: 0.02mg Dutasteride; 0.1mg Dutasteride; 0.5mg Dutasteride; Placebo
Drug: Dutasteride placebo — dutasteride placebo, by mouth once daily
  Arms: 1mg Finasteride; Placebo

SUMMARY:
The purpose of this six month study is to show that dutasteride is safe and more effective than placebo, and at least as safe and effective as finasteride in treating hair loss in men with androgenetic alopecia. Three doses of dutasteride will be investigated.

DETAILED DESCRIPTION:
Androgenetic alopecia is a common, androgen-induced, pattern of progressive loss of scalp hair with an onset at any age after puberty in genetically predisposed people. The influence of androgens on scalp hair growth is mediated by local and systemic conversion of testosterone to dihydrotestosterone , by the enzyme 5 alpha-reductase. 5 alpha-reductase has been shown to exist as 2 isoenzyme forms, Type 1 and Type 2. Type 1 is predominantly located in the skin, both in the hair follicles and sebaceous glands, and is also found in the liver and kidney . Type 2 is the dominant form in male genitalia, including the prostate, although it has also been reported to be present in the inner root sheath of the hair follicle. The presence of both isoenzymes in the hair follicles suggests that both forms are likely to be important in the pathogenesis and treatment of androgenetic alopecia. Inhibition of both Type 1 and Type 2 5 alpha-reductase may be expected to more effectively reduce systemic and local dihydrotestosterone levels than inhibition of either isoenzyme alone.

Finasteride is a selective Type 2 5 alpha-reductase inhibitor that is currently the only approved oral treatment for androgenetic alopecia worldwide. Dutasteride inhibits both Type 1 and Type 2 5alpha-reductase and is approved in more than 80 countries for the treatment of benign prostatic hyperplasia, and in Korea for the treatment of hair loss. Dutasteride is approximately 3 times as potent as finasteride at inhibiting Type 2 5 alpha-reductase and more than 100 times as potent at inhibiting Type 1 5 alpha-reductase.

In a Phase II double-blind, placebo-controlled clinical study (ARIA2004) conducted in the United States, dutasteride demonstrated significant increases in target area hair count, as compared with placebo, as early as 12 weeks. In a Phase III double- blind, placebo-controlled clinical study conducted in Korea, dutasteride 0.5 milligram (mg) demonstrated significant increases in target area hair count, as compared with placebo, at 24 weeks. This 6 month study is being conducted to provide additional evidence of the efficacy and safety of three doses of dutasteride (0.02, 0.1 and 0.5mg) in the treatment of androgenetic alopecia, and more specifically, to characterize the dose-response relationship in an ethnically-diverse population. Treatment arms will be equally balanced with approximately 180 per arm.

ELIGIBILITY:
Inclusion Criteria:

* Norwood-Hamilton Type III vertex, IV, or V

Exclusion Criteria:

* History or evidence of hair loss other than androgenetic alopecia
* Scarring of the scalp
* Use of dutasteride in previous 18 months
* Use of finasteride within previous 12 months
* Hair transplantation or hair weaving within 6 months
* Use of Minoxidil within previous 6 months
* Use of drugs with anti-androgenetic/androgenetic properties within previous 6 months
* Use of Drugs that cause hypertrichosis or hypotrichosis within previous 6 months
* Light or laser treatment of scalp within previous 3 months
* Cosmetic products aimed at improving or correcting signs of hair loss within previous 2 weeks

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 917 (Actual)
Dates: Start 2010-10-28; Primary Completion 2012-02-01 (Actual); Study Completion 2012-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (32):
- Argentina (4):
  - GSK Investigational Site, CABA, Buenos Aires
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, La Boca, Buenos Aires
  - GSK Investigational Site, Buenos Aires
- Chile (2):
  - GSK Investigational Site, Viña del Mar, Región de Valparaíso
  - GSK Investigational Site, Santiago, Región Metro de Santiago
- Japan (3):
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Tokyo
- Mexico (5):
  - GSK Investigational Site, Zapopan, Jalisco, Jalisco
  - GSK Investigational Site, Monterrey, Nuevo León
  - GSK Investigational Site, Mazatlan, Sinaloa, Sinaloa
  - GSK Investigational Site, Naucalpan, State of Mexico
  - GSK Investigational Site, Mexico City
- Peru (3):
  - GSK Investigational Site, Lima, Lima Province
  - GSK Investigational Site, Lima
  - GSK Investigational Site, Lima Cercado
- Philippines (4):
  - GSK Investigational Site, Makati City
  - GSK Investigational Site, Manila
  - GSK Investigational Site, Quezon City
  - GSK Investigational Site, Tanauan City, Batangas
- Russia (5):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Nizhny Novgorod
  - GSK Investigational Site, Ryazan
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, St'Petersburg
- Taiwan (2):
  - GSK Investigational Site, Tainan
  - GSK Investigational Site, Taipei
- Thailand (4):
  - GSK Investigational Site, Bangkoknoi Bangkok
  - GSK Investigational Site, Chiang Mai
  - GSK Investigational Site, Patumwan Bangkok
  - GSK Investigational Site, Rajthevee Bangkok

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 114263 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114263 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114263 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114263 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114263 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114263 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114263 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Dutasteride 0.02 mg: Dutasteride 0.02 milligrams (mg) and finasteride placebo once daily
- Dutasteride 0.1 mg: Dutasteride 0.1 mg and finasteride placebo once daily
- Dutasteride 0.5 mg: Dutasteride 0.5 mg and finasteride placebo once daily
- Finasteride 1 mg: Finasteride 1 mg and dutasteride placebo once daily
- Placebo: Matching dutasteride placebo and finasteride placebo once daily
Period: Overall Study
Arm/Group | Dutasteride 0.02 mg | Dutasteride 0.1 mg | Dutasteride 0.5 mg | Finasteride 1 mg | Placebo
Started | 185 | 188 | 184 | 179 | 181
Completed | 156 | 154 | 153 | 141 | 157
Not Completed | 29 | 34 | 31 | 38 | 24
Not completed — Adverse Event | 0 | 8 | 4 | 4 | 5
Not completed — Lost to Follow-up | 13 | 11 | 10 | 10 | 4
Not completed — Physician Decision | 4 | 4 | 3 | 5 | 4
Not completed — Protocol Violation | 3 | 2 | 0 | 2 | 2
Not completed — Withdrawal by Subject | 9 | 9 | 14 | 17 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dutasteride 0.02 mg | Dutasteride 0.1 mg | Dutasteride 0.5 mg | Finasteride 1 mg | Placebo | Total
Number analyzed (Participants) | 185 | 188 | 184 | 179 | 181 | 917
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.5 (7.72) | 38.7 (7.44) | 38.6 (7.66) | 38.0 (7.81) | 38.7 (8.43) | 38.5 (7.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 185 | 188 | 184 | 179 | 181 | 917
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian - Japanese Heritage | 40 | 40 | 40 | 40 | 39 | 199
  American Indian or Alaskan Native | 37 | 38 | 39 | 36 | 38 | 188
  African American/African Heritage | 1 | 0 | 0 | 0 | 1 | 2
  Asian - South East Asian Heritage | 44 | 43 | 42 | 41 | 41 | 211
  Asian - East Asian Heritage | 19 | 20 | 19 | 19 | 19 | 96
  Asian - Mixed Race | 0 | 0 | 0 | 0 | 1 | 1
  White - White/Caucasian/European Heritage | 44 | 47 | 44 | 43 | 42 | 220

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (BL) in Target Area Hair Count (HC) Within a 2.54 Centimeter (cm) (1 Inch) Diameter Circle at the Vertex at Week 24, as Assessed by Macrophotographic Technique (MT)
Description: The primary target area HC was based on the nonvellus hair (>=30 micrometers [μm] in width; thick and noticeable hair) count within a target 2.54 cm (1 inch) diameter circle at the vertex (crown, topmost part of the head). A cosmetic ink dot was placed by tattoo at BL so that the same area could be identified at BL and post-BL. If the ink dot faded, it was re-done in exactly the same location to ensure visibility for subsequent photographs. For the MT, hair was clipped before each photograph; HC was based on hair follicles in the photographs. Change from BL=Week 24 value minus the BL value.
Time Frame: Baseline and Week 24
Population: Intent-to-Treat (ITT) Population: all randomized participants regardless of whether or not treatment was administered. Calculation was based on the last observation carried forward (LOCF) imputation method for missing data. All participants for whom data were collected at both Baseline and Week 24 were assessed.
Measure: Least Squares Mean (Standard Error); unit: Hair count
Groups:
- Placebo: Matching dutasteride placebo and finasteride placebo once daily by mouth for 24 weeks (6 months). Placebo treatment was taken either with or without food.
- Dutasteride 0.02 mg: Dutasteride 0.02 milligrams (mg) and finasteride placebo once daily by mouth for 24 weeks (6 months). Study treatment was taken either with or without food.
- Dutasteride 0.1 mg: Dutasteride 0.1 mg and finasteride placebo once daily by mouth for 24 weeks (6 months). Study treatment was taken either with or without food.
- Dutasteride 0.5 mg: Dutasteride 0.5 mg and finasteride placebo once daily by mouth for 24 weeks (6 months). Study treatment was taken either with or without food.
- Finasteride 1 mg: Finasteride 1 mg and dutasteride placebo once daily by mouth for 24 weeks (6 months). Active comparator was taken either with or without food.
Arm/Group | Placebo | Dutasteride 0.02 mg | Dutasteride 0.1 mg | Dutasteride 0.5 mg | Finasteride 1 mg
Number analyzed (Participants) | 148 | 155 | 158 | 150 | 141
Hair count | -4.9 (7.89) | 17.1 (7.74) | 63.0 (7.67) | 89.6 (7.87) | 56.5 (8.12)
Statistical Analysis 1: Comparison: Placebo vs Dutasteride 0.02 mg; Test type: Superiority or Other; p = 0.046, General linear model; Least-squares (LS) mean difference = 22, 98.33% CI 2-sided [-4.4 to 48.4] — Estimates are based on the adjusted (least-squares) means from the general linear model: Change from Baseline = Treatment + Cluster + Baseline Value. The estimation value represents the dutasteride 0.02 mg LS mean minus the placebo LS mean
Statistical Analysis 2: Comparison: Placebo vs Dutasteride 0.1 mg; Test type: Superiority or Other; p < 0.001, General linear model; LS mean difference = 67.9, 98.33% CI 2-sided [41.6 to 94.2] — Estimates are based on the adjusted (least-squares) means from the general linear model: Change from Baseline = Treatment + Cluster + Baseline Value. The estimation value represents the dutasteride 0.1 mg LS mean minus the placebo LS mean
Statistical Analysis 3: Comparison: Placebo vs Dutasteride 0.5 mg; Test type: Superiority or Other; p < 0.001, General linear model; Each dose of dutasteride independently analyzed for comparison against placebo using a general linear model; LS mean difference = 94.4, 98.33% CI 2-sided [67.8 to 121.0] — Estimates are based on the adjusted (least-squares) means from the general linear model: Change from Baseline = Treatment + Cluster + Baseline Value. The estimation value represents the dutasteride 0.5 mg LS mean minus the placebo LS mean
Statistical Analysis 4: Comparison: Placebo vs Finasteride 1 mg; Test type: Superiority or Other; p < 0.001, General linear model; Least squares mean difference = 61.4, 98.33% CI 2-sided [34.4 to 88.4] — Estimates are based on the adjusted (least-squares) means from the general linear model: Change from Baseline = Treatment + Cluster + Baseline Value. The estimation value represents the finasteride 1 mg LS mean minus the placebo LS mean
Statistical Analysis 5: Comparison: Dutasteride 0.02 mg vs Finasteride 1 mg; Test type: Non-Inferiority or Equivalence — Differences between dutasteride (DUT) and finasteride (FIN) were assessed using a general linear model (GLM) adjusted for treatment, cluster, and BL hair count (HC). The one-sided 99.165% confidence interval (CI) for DUT minus FIN was derived, and noninferiority (NI) demonstrated if the lower end of the CI was greater than -35 hairs. If NI was achieved with a dose of DUT, the primary endpoint was to be analyzed for superiority against FIN using a GLM adjusted for treatment, cluster, and BL HC; p < 0.001, General linear model; Least squares mean difference = -39.4, 99.165% CI [-66.1 to -12.7] — Estimates are based on the adjusted (least-squares) means from the general linear model: Change from Baseline = Treatment + Cluster + Baseline Value. The estimation value represents the finasteride 1 mg LS mean minus the Dutasteride 0.02 mg LS mean
Statistical Analysis 6: Comparison: Dutasteride 0.1 mg vs Finasteride 1 mg; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 5]; p = 0.28, General linear model; Least squares mean difference = 6.5, 99.165% CI [-20.1 to 33.1] — Estimates are based on the adjusted (least-squares) means from the general linear model: Change from Baseline = Treatment + Cluster + Baseline Value. The estimation value represents the finasteride 1 mg LS mean minus the Dutasteride 0.1 mg LS mean
Statistical Analysis 7: Comparison: Dutasteride 0.5 mg vs Finasteride 1 mg; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 5]; p = 0.002, General linear model; Least squares mean difference = 33, 99.165% CI [6.1 to 60] — Estimates are based on the adjusted (least-squares) means from the general linear model: Change from Baseline = Treatment + Cluster + Baseline Value. The estimation value represents the finasteride 1 mg LS mean minus the Dutasteride 0.5 mg LS mean
Statistical Analysis 8: Comparison: Dutasteride 0.02 mg vs Finasteride 1 mg; Test type: Superiority or Other; p < 0.001, General linear model; Least squares mean difference = -39.4, 98.33% CI 2-sided [-66.1 to -12.7] — [estimate comment as in outcome 1, analysis 5]
Statistical Analysis 9: Comparison: Dutasteride 0.1 mg vs Finasteride 1 mg; Test type: Superiority or Other; p = 0.56, General linear model; Least squares mean difference = 6.5, 98.33% CI 2-sided [-20.1 to 33.1] — [estimate comment as in outcome 1, analysis 6]
Statistical Analysis 10: Comparison: Dutasteride 0.5 mg vs Finasteride 1 mg; Test type: Superiority or Other; p = 0.003, General linear model; Least squares mean difference = 33, 98.33% CI 2-sided [6.1 to 60] — [estimate comment as in outcome 1, analysis 7]

2. Secondary Outcome: Change From Baseline in Target Area Hair Count Within a 1.13 cm (0.44 Inch) Diameter Circle at the Vertex at Week 24, as Assessed by MT
Description: The primary target area HC was based on the nonvellus hair (>=30 micrometers [μm] in width; thick and noticeable hair) count within a target 1.13 cm (0.44 inch) diameter circle at the vertex (crown, topmost part of the head). A cosmetic ink dot was placed by tattoo at BL so that the same area could be identified at BL and post-BL. If the ink dot faded, it was re-done in exactly the same location to ensure visibility for subsequent photographs. For the MT, hair was clipped before each photograph; HC was based on hair follicles in the photographs. Change from BL=Week 24 value minus the BL value.
Time Frame: Baseline and Week 24
Population: ITT Population. Calculation was based on the LOCF imputation method for missing data. All participants for whom data were collected at both Baseline and Week 24 were assessed.
Measure: Least Squares Mean (Standard Error); unit: Hair count
Arm/Group | Placebo | Dutasteride 0.02 mg | Dutasteride 0.1 mg | Dutasteride 0.5 mg | Finasteride 1 mg
Number analyzed (Participants) | 152 | 158 | 159 | 152 | 142
Hair count | -0.3 (1.74) | 4.2 (1.71) | 12.4 (1.70) | 18.1 (1.74) | 12.1 (1.80)

3. Secondary Outcome: Change From Baseline in Target Area Hair Count Within a 2.54 cm (1 Inch) Diameter Circle at the Vertex at Week 12 as Assessed by MT
Description: The primary target area HC was based on the nonvellus hair (>=30 micrometers [μm] in width; thick and noticeable hair) count within a target 2.54 cm (1 inch) diameter circle at the vertex (crown, topmost part of the head). A cosmetic ink dot was placed by tattoo at BL so that the same area could be identified at BL and post-BL. If the ink dot faded, it was re-done in exactly the same location to ensure visibility for subsequent photographs. For the MT, hair was clipped before each photograph; HC was based on hair follicles in the photographs. Change from BL=Week 12 value minus the BL value.
Time Frame: Baseline and Week 12
Population: ITT Population. Calculation was based on the LOCF imputation method for missing data. All participants for whom data were collected at both Baseline and Week 12 were assessed.
Measure: Least Squares Mean (Standard Error); unit: Hair count
Arm/Group | Placebo | Dutasteride 0.02 mg | Dutasteride 0.1 mg | Dutasteride 0.5 mg | Finasteride 1 mg
Number analyzed (Participants) | 147 | 144 | 151 | 145 | 131
Hair count | -4.0 (7.22) | 22.9 (7.32) | 59.6 (7.15) | 82.3 (7.29) | 50.9 (7.67)

4. Secondary Outcome: Change From Baseline in Target Area Hair Count Within a 1.13 cm (0.44 Inch) Diameter Circle at the Vertex, as Assessed by MT at Week 12
Description: The primary target area HC was based on the nonvellus hair (>=30 micrometers [μm] in width; thick and noticeable hair) count within a target 1.13 cm (0.44 inch) diameter circle at the vertex (crown, topmost part of the head). A cosmetic ink dot was placed by tattoo at BL so that the same area could be identified at BL and post-BL. If the ink dot faded, it was re-done in exactly the same location to ensure visibility for subsequent photographs. For the MT, hair was clipped before each photograph; HC was based on hair follicles in the photographs. Change from BL=Week 12 value minus the BL value.
Time Frame: Baseline and Week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Hair count
Arm/Group | Placebo | Dutasteride 0.02 mg | Dutasteride 0.1 mg | Dutasteride 0.5 mg | Finasteride 1 mg
Number analyzed (Participants) | 152 | 154 | 155 | 149 | 134
Hair count | -0.4 (1.63) | 5.1 (1.63) | 12.8 (1.62) | 17.1 (1.65) | 10.8 (1.74)

5. Secondary Outcome: Change From Baseline in Target Area Hair Width Within a 2.54 cm (1 Inch) Diameter Circle at the Vertex at Week 12 and Week 24, as Assessed by MT
Description: The target area hair width was the sum of all nonvellus hairs (>=30 µm in width; thick and noticeable hair) within a target 2.54 cm (1 inch) diameter circle at the vertex (crown, topmost part of the head). For the MT, hair was clipped before each photograph. A cosmetic ink dot was placed by tattoo at Baseline so that the same area could be identified at Baseline and post-Baseline. If the ink dot faded, it was re-done in exactly the same location to ensure it was visible for subsequent photographs. Change from Baseline was calculated as the Week 12 or Week 24 value minus the Baseline value.
Time Frame: Baseline, Week 12, and Week 24
Population: ITT Population. Calculation was based on the LOCF imputation method for missing data. All participants for whom data were collected at Baseline, Week 12, and Week 24 were assessed.
Measure: Least Squares Mean (Standard Error); unit: millimeters
Arm/Group | Placebo | Dutasteride 0.02 mg | Dutasteride 0.1 mg | Dutasteride 0.5 mg | Finasteride 1 mg
Number analyzed (Participants) | 148 | 155 | 158 | 150 | 141
millimeters
  Week 12, n=147, 144, 151, 145, 131 | -0.7 (0.40) | 0.3 (0.41) | 3.1 (0.40) | 4.7 (0.41) | 3.2 (0.43)
  Week 24, n=148, 155, 158, 150, 141 | -0.9 (0.45) | -0.0 (0.44) | 3.9 (0.44) | 5.8 (0.45) | 4.0 (0.46)

6. Secondary Outcome: Change From Baseline in Target Area Hair Width Within a 1.13 cm (0.44 Inch) Diameter Circle at the Vertex at Week 12 and Week 24, as Assessed by MT
Description: The target area hair width was the sum of all nonvellus hairs (>=30 µm in width; thick and noticeable hair) within a target 1.13 cm (0.44 inch) diameter circle at the vertex (crown, topmost part of the head). For the MT, hair was clipped before each photograph. A cosmetic ink dot was placed by tattoo at Baseline so that the same area could be identified at Baseline and post-Baseline. If the ink dot faded, it was re-done in exactly the same location to ensure it was visible for subsequent photographs. Change from Baseline was calculated as the Week 12 or Week 24 value minus the Baseline value.
Time Frame: Baseline, Week 12, and Week 24
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: millimeters
Arm/Group | Placebo | Dutasteride 0.02 mg | Dutasteride 0.1 mg | Dutasteride 0.5 mg | Finasteride 1 mg
Number analyzed (Participants) | 152 | 158 | 159 | 152 | 142
millimeters
  Week 12, n=152, 154, 155, 149, 134 | -0.1 (0.09) | 0.1 (0.09) | 0.7 (0.09) | 0.9 (0.09) | 0.6 (0.10)
  Week 24, n=152, 158, 159, 152, 142 | -0.2 (0.10) | 0.1 (0.10) | 0.8 (0.10) | 1.2 (0.10) | 0.8 (0.10)

7. Secondary Outcome: Change From Baseline in Terminal Hair Count (THC) Within a 2.54 cm (1 Inch) Diameter Circle at the Vertex at Week 12 and Week 24, as Assessed by MT
Description: The THC (thick, long, and dark hair) was the sum of all nonvellus hairs (>=60 μm in width; thick and noticeable hair) within a target 2.54 cm (1 inch) diameter circle at the vertex (crown, topmost part of the head). A cosmetic ink dot was placed by tattoo at BL so that the same area could be identified at BL and post-BL. If the ink dot faded, it was re-done in exactly the same location to ensure visibility for subsequent photographs. For the MT, hair was clipped before each photograph; HC was based on the hair follicles in the photographs. Change from BL=Week 12/Week 24 value minus BL value.
Time Frame: Baseline, Week 12, and Week 24
Population: ITT Population. Calculation was based on the LOCF imputation method for missing data. All participants for whom data were collected at both Baseline, Week 12, and Week 24 were assessed.
Measure: Least Squares Mean (Standard Error); unit: Hair count
Arm/Group | Placebo | Dutasteride 0.02 mg | Dutasteride 0.1 mg | Dutasteride 0.5 mg | Finasteride 1 mg
Number analyzed (Participants) | 148 | 155 | 158 | 150 | 141
Hair count
  Week 12, n=147, 144, 151, 145, 131 | -11.5 (4.39) | -13.4 (4.44) | 18.3 (4.35) | 29.3 (4.43) | 24.2 (4.67)
  Week 24, n=148, 155, 158, 150, 141 | -17.5 (5.13) | -15.7 (5.03) | 29.4 (4.99) | 46 (5.11) | 36.3 (5.28)

8. Secondary Outcome: Change From Baseline in Terminal Hair Count Within a 1.13 cm (0.44 Inch) Diameter Circle at the Vertex at Week 12 and Week 24, as Assessed by MT
Description: The THC (thick, long, and dark hair) was the sum of all nonvellus hairs (>=60 μm in width; thick and noticeable hair) within a target 1.13 cm (0.44 inch) diameter circle at the vertex (crown, topmost part of the head). A cosmetic ink dot was placed by tattoo at BL so that the same area could be identified at BL and post-BL. If the ink dot faded, it was re-done in exactly the same location to ensure visibility for subsequent photographs. For the MT, hair was clipped before each photograph; HC was based on hair follicles in the photographs. Change from BL=Week 12/Week 24 value minus BL value.
Time Frame: Baseline, Week 12, and Week 24
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: Hair count
Arm/Group | Placebo | Dutasteride 0.02 mg | Dutasteride 0.1 mg | Dutasteride 0.5 mg | Finasteride 1 mg
Number analyzed (Participants) | 152 | 158 | 159 | 152 | 142
Hair count
  Week 12, n=152, 154, 155, 149, 134 | -1.1 (1.05) | -2.7 (1.05) | 4.0 (1.05) | 5.9 (1.06) | 4.5 (1.12)
  Week 24, n=152, 158, 159, 152, 142 | -3.0 (1.20) | -2.8 (1.18) | 6.0 (1.18) | 9.3 (1.20) | 7.2 (1.25)

9. Secondary Outcome: Global Assessment of Improvement From Baseline to Week 24 Assessed for Vertex and Frontal Views Separately
Description: A central panel of 3 dermatologists independently assessed change in hair growth from Baseline to Week 24 using a 7-point scale: greatly decreased (-3), moderately decreased (-2), slightly decreased (-1), no change (0), slightly increased (1), moderately increased (2), and greatly increased (3). The median score, across the 3 panel members, is summarized. This assessment was performed by comparing the global photographs obtained at Baseline with those subsequently obtained at Week 24. This assessment was made separately based on the global photography of the vertex and frontal views.
Time Frame: Baseline and Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Dutasteride 0.02 mg | Dutasteride 0.1 mg | Dutasteride 0.5 mg | Finasteride 1 mg
Number analyzed (Participants) | 172 | 174 | 176 | 167 | 165
scores on a scale
  Vertex view, n=172, 174, 176, 167, 164 | -0.15 (0.056) | -0.09 (0.056) | 0.42 (0.055) | 0.63 (0.057) | 0.49 (0.057)
  Frontal/Superior view, n=171, 174, 176, 167, 165 | -0.14 (0.054) | -0.10 (0.053) | 0.36 (0.053) | 0.58 (0.055) | 0.34 (0.055)

10. Secondary Outcome: Change From Baseline in Investigator Photographic Assessment Questionnaire (IPAQ) Scores Assessed at Week 12 for Vertex and Frontal Views Separately
Description: The IPAQ was completed by the Investigator or designee by comparing the global photographs obtained at Baseline with those obtained at Week 12. This assessment was made separately based on the global photography of the vertex and frontal views. The change from Baseline in hair growth was assessed using the following 7-point scale: -3 = greatly decreased, -2 = moderately decreased, -1 = slightly decreased, 0 = no change, +1 = slightly increased, +2 = moderately increased, +3 = greatly increased.
Time Frame: Baseline and Week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Dutasteride 0.02 mg | Dutasteride 0.1 mg | Dutasteride 0.5 mg | Finasteride 1 mg
Number analyzed (Participants) | 172 | 171 | 172 | 166 | 160
scores on a scale
  Vertex view | 0.48 (0.068) | 0.35 (0.069) | 0.62 (0.068) | 0.78 (0.070) | 0.70 (0.071)
  Frontal view | 0.30 (0.059) | 0.33 (0.059) | 0.54 (0.059) | 0.55 (0.060) | 0.55 (0.061)

11. Secondary Outcome: Change From Baseline in Investigator Photographic Assessment Questionnaire (IPAQ) Scores Assessed at Week 24 for Vertex and Frontal Views Separately
Description: as for outcome 10
Time Frame: Baseline and Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Dutasteride 0.02 mg | Dutasteride 0.1 mg | Dutasteride 0.5 mg | Finasteride 1 mg
Number analyzed (Participants) | 173 | 174 | 177 | 167 | 165
scores on a scale
  Vertex view | 0.36 (0.079) | 0.37 (0.079) | 1.03 (0.078) | 1.30 (0.080) | 1.07 (0.081)
  Frontal view | 0.30 (0.075) | 0.28 (0.075) | 0.78 (0.074) | 1.11 (0.076) | 0.88 (0.077)

12. Secondary Outcome: Number of Participants With the Indicated Change From Baseline (BL) in the Stage (S) of Androgenic Alopecia (AGA) According to the Norwood-Hamilton Scale at Week 12 (W12)
Description: The investigator/designee assessed the stage (Stage I to Stage VII) of AGA (i.e., male pattern baldness [MPB]) by utilizing the Norwood-Hamilton scale, used to measure the progression of MPB. Stage VII indicates worse balding than stage I. Assessment was made by direct visual examination (aided by pictures) of the participant at Baseline and Week 12 (W12). "v," vertex; most of the hair loss (commonly seen with advancing age) is on the vertex. "a," type a variant; major features are (1) the entire anterior hairline border recedes in unison; (2) there is no simultaneous balding of the vertex.
Time Frame: Baseline and Week 12
Population: ITT Population. Calculation was based on the LOCF imputation method for missing data. All participants for whom data were collected at both Baseline and Week 12 were assessed. The number of participants analyzed reflects the sum of the participants with the three BL stages.
Measure: Number; unit: participants
Arm/Group | Placebo | Dutasteride 0.02 mg | Dutasteride 0.1 mg | Dutasteride 0.5 mg | Finasteride 1 mg
Number analyzed (Participants) | 172 | 177 | 173 | 169 | 161
participants
  BL S IIIv to W12 S II, n=79, 70, 69, 72, 73 | 1 | 1 | 0 | 1 | 0
  BL S IIIv to W12 S IIa, n=79, 70, 69, 72, 73 | 0 | 0 | 0 | 0 | 0
  BL S IIIv to W12 S III, n=79, 70, 69, 72, 73 | 4 | 8 | 11 | 10 | 11
  BL S IIIv to W12 S IIIa, n=79, 70, 69, 72, 73 | 0 | 0 | 1 | 0 | 0
  BL S IIIv to W12 S IIIv, n=79, 70, 69, 72, 73 | 71 | 59 | 55 | 59 | 62
  BL S IIIv to W12 S IV, n=79, 70, 69, 72, 73 | 2 | 1 | 2 | 2 | 0
  BL S IIIv to W12 S IVa, n=79, 70, 69, 72, 73 | 0 | 0 | 0 | 0 | 0
  BL S IIIv to W12 S V, n=79, 70, 69, 72, 73 | 1 | 1 | 0 | 0 | 0
  BL S IIIv to W12 S Va, n=79, 70, 69, 72, 73 | 0 | 0 | 0 | 0 | 0
  BL S IIIv to W12 S VI, n=79, 70, 69, 72, 73 | 0 | 0 | 0 | 0 | 0
  BL S IV to W12 S II, n=52, 59, 58, 56, 53 | 0 | 0 | 0 | 0 | 0
  BL S IV to W12 S IIa, n=52, 59, 58, 56, 53 | 0 | 0 | 0 | 0 | 0
  BL S IV to W12 S III, n=52, 59, 58, 56, 53 | 2 | 4 | 1 | 4 | 1
  BL S IV to W12 S IIIa, n=52, 59, 58, 56, 53 | 0 | 0 | 0 | 0 | 0
  BL S IV to W12 S IIIv, n=52, 59, 58, 56, 53 | 2 | 3 | 8 | 5 | 5
  BL S IV to W12 S IV, n=52, 59, 58, 56, 53 | 45 | 50 | 44 | 47 | 45
  BL S IV to W12 S IVa, n=52, 59, 58, 56, 53 | 1 | 0 | 1 | 0 | 0
  BL S IV to W12 S V, n=52, 59, 58, 56, 53 | 2 | 2 | 4 | 0 | 2
  BL S IV to W12 S Va, n=52, 59, 58, 56, 53 | 0 | 0 | 0 | 0 | 0
  BL S IV to W12 S VI, n=52, 59, 58, 56, 53 | 0 | 0 | 0 | 0 | 0
  BL S V to W12 S II, n=41, 46, 46, 41, 35 | 0 | 0 | 0 | 0 | 0
  BL S V to W12 S IIa, n=41, 46, 46, 41, 35 | 0 | 0 | 0 | 0 | 0
  BL S V to W12 S III, n=41, 46, 46, 41, 35 | 2 | 1 | 0 | 1 | 0
  BL S V to W12 S IIIa, n=41, 46, 46, 41, 35 | 0 | 0 | 0 | 0 | 0
  BL S V to W12 S IIIv, n=41, 46, 46, 41, 35 | 0 | 1 | 3 | 1 | 0
  BL S V to W12 S IV, n=41, 46, 46, 41, 35 | 4 | 4 | 5 | 5 | 2
  BL S V to W12 S IVa, n=41, 46, 46, 41, 35 | 0 | 0 | 0 | 0 | 0
  BL S V to W12 S V, n=41, 46, 46, 41, 35 | 35 | 40 | 38 | 33 | 33
  BL S V to W12 S Va, n=41, 46, 46, 41, 35 | 0 | 0 | 0 | 0 | 0
  BL S V to W12 S VI, n=41, 46, 46, 41, 35 | 0 | 0 | 0 | 1 | 0

13. Secondary Outcome: Number of Participants With the Indicated Change From Baseline (BL) in the Stage (S) of Androgenic Alopecia (AGA) According to the Norwood-Hamilton Scale at Week 24
Description: The investigator/designee assessed the stage (Stage I to Stage VII) of AGA (i.e., male pattern baldness [MPB]) by utilizing the Norwood-Hamilton scale, used to measure the progression of MPB. Stage VII indicates worse balding than stage I. Assessment was made by direct visual examination (aided by pictures) of the participant at Baseline and Week 24 (W24). "v," vertex; most of the hair loss (commonly seen with advancing age) is on the vertex. "a," type a variant; major features are (1) the entire anterior hairline border recedes in unison; (2) there is no simultaneous balding of the vertex.
Time Frame: Baseline and Week 24
Population: ITT Population. Calculation was based on the LOCF imputation method for missing data. All participants for whom data were collected at both Baseline and Week 24 were assessed. The number of participants analyzed reflects the sum of the participants with the three BL stages.
Measure: Number; unit: participants
Arm/Group | Placebo | Dutasteride 0.02 mg | Dutasteride 0.1 mg | Dutasteride 0.5 mg | Finasteride 1 mg
Number analyzed (Participants) | 173 | 177 | 177 | 169 | 165
participants
  BL S IIIv to W24 S II, n=80, 72, 72, 72, 76 | 3 | 2 | 2 | 3 | 2
  BL S IIIv to W24 S IIa, n=80, 72, 72, 72, 76 | 0 | 0 | 0 | 1 | 1
  BL S IIIv to W24 S III, n=80, 72, 72, 72, 76 | 6 | 8 | 11 | 13 | 13
  BL S IIIv to W24 S IIIa, n=80, 72, 72, 72, 76 | 0 | 0 | 0 | 0 | 0
  BL S IIIv to W24 S IIIv, n=80, 72, 72, 72, 76 | 67 | 61 | 58 | 54 | 59
  BL S IIIv to W24 S IV, n=80, 72, 72, 72, 76 | 4 | 1 | 1 | 1 | 1
  BL S IIIv to W24 S IVa, n=80, 72, 72, 72, 76 | 0 | 0 | 0 | 0 | 0
  BL S IIIv to W24 S V, n=80, 72, 72, 72, 76 | 0 | 0 | 0 | 0 | 0
  BL S IIIv to W24 S Va, n=80, 72, 72, 72, 76 | 0 | 0 | 0 | 0 | 0
  BL S IIIv to W24 S VI, n=80, 72, 72, 72, 76 | 0 | 0 | 0 | 0 | 0
  BL S IV to W24 S II, n=52, 59, 59, 56, 54 | 0 | 1 | 1 | 1 | 0
  BL S IV to W24 S IIa, n=52, 59, 59, 56, 54 | 0 | 0 | 0 | 0 | 0
  BL S IV to W24 S III, n=52, 59, 59, 56, 54 | 2 | 3 | 4 | 5 | 4
  BL S IV to W24 S IIIa, n=52, 59, 59, 56, 54 | 0 | 0 | 0 | 2 | 0
  BL S IV to W24 S IIIv, n=52, 59, 59, 56, 54 | 4 | 7 | 11 | 10 | 13
  BL S IV to W24 S IV, n=52, 59, 59, 56, 54 | 44 | 46 | 39 | 37 | 36
  BL S IV to W24 S IVa, n=52, 59, 59, 56, 54 | 0 | 0 | 0 | 1 | 0
  BL S IV to W24 S V, n=52, 59, 59, 56, 54 | 2 | 2 | 4 | 0 | 1
  BL S IV to W24 S Va, n=52, 59, 59, 56, 54 | 0 | 0 | 0 | 0 | 0
  BL S IV to W24 S VI, n=52, 59, 59, 56, 54 | 0 | 0 | 0 | 0 | 0
  BL S V to W24 S II, n=41, 46, 46, 41, 35 | 0 | 1 | 0 | 0 | 0
  BL S V to W12 S IIa, n=41, 46, 46, 41, 35 | 0 | 0 | 0 | 0 | 0
  BL S V to W24 S III, n=41, 46, 46, 41, 35 | 2 | 1 | 1 | 3 | 1
  BL S V to W24 S IIIa, n=41, 46, 46, 41, 35 | 0 | 0 | 0 | 0 | 0
  BL S V to W24 S IIIv, n=41, 46, 46, 41, 35 | 3 | 1 | 4 | 3 | 1
  BL S V to W24 S IV, n=41, 46, 46, 41, 35 | 7 | 10 | 8 | 10 | 8
  BL S V to W24 S IVa, n=41, 46, 46, 41, 35 | 0 | 0 | 0 | 0 | 1
  BL S V to W24 S V, n=41, 46, 46, 41, 35 | 29 | 33 | 33 | 25 | 24
  BL S V to W24 S Va, n=41, 46, 46, 41, 35 | 0 | 0 | 0 | 0 | 0
  BL S V to W24 S VI, n=41, 46, 46, 41, 35 | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Serum Concentration of Dutasteride at Week 12, Week 24, and Follow-up (Week 26)
Description: Serum concentrations of dutasteride were measured after 12 weeks and 24 weeks of study treatment and at follow-up (approximately 2 weeks after the last dose of study treatment).
Time Frame: Week 12, Week 24, and Week 26
Population: ITT Population. All participants for whom data were collected at Baseline, Week 12, and Week 24 were assessed.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Dutasteride 0.02 mg | Dutasteride 0.1 mg | Dutasteride 0.5 mg
Number analyzed (Participants) | 172 | 172 | 165
nanograms per milliliter (ng/mL)
  Week 12, n=172, 172, 165 | 0.2 (1.96) | 2.1 (1.72) | 33.2 (20.10)
  Week 24, n=158, 158, 153 | 0.0 (0.14) | 2.0 (1.90) | 36.1 (23.21)
  Week 26, n=156, 154, 152 | 0.1 (0.84) | 0.3 (0.69) | 21.1 (17.65)

15. Secondary Outcome: Serum Dihydrotestosterone (DHT) at Week 12, Week 24, and Follow-up (Week 26)
Description: Serum concentrations of DHT were measured after 12 weeks and 24 weeks of study treatment and at follow-up (approximately 2 weeks after the last dose of study treatment).
Time Frame: Week 12, Week 24, and Week 26
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: nanomoles per liter (nmol/L)
Arm/Group | Placebo | Dutasteride 0.02 mg | Dutasteride 0.1 mg | Dutasteride 0.5 mg | Finasteride 1 mg
Number analyzed (Participants) | 173 | 177 | 177 | 171 | 165
nanomoles per liter (nmol/L)
  Week 12, n=172, 174, 172, 170, 161 | 1.17 (0.531) | 0.88 (0.519) | 0.39 (0.402) | 0.31 (0.374) | 0.45 (0.462)
  Week 24, n=173, 177, 176, 170, 165 | 1.16 (0.482) | 1.01 (0.540) | 0.49 (0.500) | 0.31 (0.402) | 0.49 (0.500)
  Week 26, n=173, 177, 177, 171, 165 | 1.21 (0.523) | 1.11 (0.600) | 0.77 (0.602) | 0.37 (0.451) | 1.03 (0.636)

16. Secondary Outcome: Change From Baseline in Hair Growth Index (HGI) Scores at Weeks 12 and 24
Description: Participant-perceived change in HG was assessed by 3 questions (each scored on a 7-point scale) on a health outcome questionnaire: "Since the start of treatment, when I look at my thinning area, I can see...", "Since the start of treatment, my hair now covers…", and "Since the start of treatment, the appearance (thickness/quality/amount) of the thinning area on my head is…" -3, Much less; -2, Moderately less; -1, Slightly less; 0, The same amount; 1, Slightly more; 2, Moderately more; 3, Much more scalp. The scores for the 3 questions were summed to obtain the HGI total score (-9 to 9).
Time Frame: Baseline, Week 12, and Week 24
Population: ITT Population. Calculation was based on the LOCF imputation method for missing data. All participants for whom data were collected at Week 12 and Week 24 were assessed.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Dutasteride 0.02 mg | Dutasteride 0.1 mg | Dutasteride 0.5 mg | Finasteride 1 mg
Number analyzed (Participants) | 172 | 174 | 177 | 167 | 165
scores on a scale
  Week 12, n=171, 171, 172, 166, 160 | 1.2 (0.19) | 0.9 (0.19) | 1.7 (0.19) | 2.0 (0.19) | 1.7 (0.20)
  Week 24, n=172, 174, 177, 167, 165 | 1.1 (0.22) | 1.1 (0.22) | 2.8 (0.22) | 3.2 (0.22) | 2.5 (0.23)

17. Secondary Outcome: Change From Baseline in Total Hair Growth Satisfaction Scale (HGSS) Scores at Weeks 12 and 24
Description: Participant satisfaction with hair appearance/growth was assessed by 5 questions (each scored on a 7-point scale: How satisfied do you feel about: [1] The overall appearance of your hair; [2] The appearance of the thinning area[s] [TAs] on your head; [3] The amount of scalp that can be seen in the TAs; [4] The amount of hair in the TAs; [5] The growth of hair in the TAs): -3, Very dissatisfied (DS); -2, DS; -1, Somewhat DS; 0, Neutral (neither satisfied nor DS); 1, Somewhat satisfied (SA); 2, SA; 3, Very SA. The scores for the 5 questions were summed to obtain the HGSS total score (-15 to 15).
Time Frame: Baseline, Week 12, and Week 24
Population: as for outcome 16
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Dutasteride 0.02 mg | Dutasteride 0.1 mg | Dutasteride 0.5 mg | Finasteride 1 mg
Number analyzed (Participants) | 172 | 176 | 177 | 170 | 165
scores on a scale
  Week 12, n=171, 174, 173, 170, 160 | 8.5 (0.54) | 7.9 (0.53) | 9.8 (0.53) | 8.4 (0.54) | 8.5 (0.55)
  Week 24, n=172, 176, 177, 170, 165 | 9.3 (0.56) | 8.3 (0.56) | 11.5 (0.56) | 12.5 (0.56) | 10.8 (0.59)

ADVERSE EVENTS:
Arm/Group | Dutasteride 0.02 mg | Dutasteride 0.1 mg | Dutasteride 0.5 mg | Finasteride 1 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/185 | 3/188 | 1/184 | 2/179 | 2/181
Other Adverse Events (participants affected / at risk) | 34/185 | 34/188 | 41/184 | 32/179 | 36/181
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dutasteride 0.02 mg (N=185) | Dutasteride 0.1 mg (N=188) | Dutasteride 0.5 mg (N=184) | Finasteride 1 mg (N=179) | Placebo (N=181)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cartilage injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fractured sacrum (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection parasitic (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngeal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Salmonellosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dutasteride 0.02 mg (N=185) | Dutasteride 0.1 mg (N=188) | Dutasteride 0.5 mg (N=184) | Finasteride 1 mg (N=179) | Placebo (N=181)
Erectile dysfunction (Reproductive system and breast disorders) | 8 | 7 | 10 | 10 | 7
Headache (Nervous system disorders) | 8 | 8 | 11 | 5 | 16
Libido decreased (Psychiatric disorders) | 10 | 9 | 6 | 9 | 2
Nasopharyngitis (Infections and infestations) | 19 | 15 | 23 | 14 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.